CLINICAL TRIAL: NCT03302273
Title: Topical Cadaveric-Derived Corneal Epithelial Stem Cell Transplant Therapy for the Treatment of Severe Dry Eye Disease
Brief Title: Corneal Epithelial Stem Cells and Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sloan W. Rush, MD (Other)
Responsible Party: Sponsor-Investigator, Sloan W. Rush, MD, Physician, Panhandle Eye Group, LLP
Organization: Panhandle Eye Group, LLP (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2017-09-30; First posted 2017-10-05 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes; Dry Eye; Ocular Inflammation; Ocular Surface Disease; Ocular Discomfort; Blepharitis
Keywords: stem cell therapy; dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes; Blepharitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal Epithelial Stem Cell Transplant (Experimental): The treatment will consist of transplantation (via self-administration) of formulated topical eye drops containing cadaveric epithelial stem cell-derived biologic material four times daily in both eyes for a three month interval.
  Interventions: Other: Corneal Epithelial Stem Cell Transplant

INTERVENTIONS:
Other: Corneal Epithelial Stem Cell Transplant — Self-administration of formulated topical eye drops containing cadaveric epithelial stem cell-derived biologic material.

SUMMARY:
To study of a novel, therapeutic Human Cells, Tissues, and Cellular and Tissue-Based Product (HCT/P) in the treatment of severe dry eye disease that is failing conventional treatments. This pilot study will carefully observe and monitor each qualifying and willing individual for response to treatment, signs of toxicity and adverse effects from the treatment, and for ability of the treatment to improve comfort and restore vision.

DETAILED DESCRIPTION:
Eligible patients presenting with severe dry eye disease that have failed treatment with conventional measures will be screened for inclusion into the study. The treatment will consist of administration of formulated topical eye drops containing cadaveric epithelial stem cell-derived product. These eye drops will be transplanted by topical self-administration by the patient four times daily in both eyes for a three month interval.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced dry eye disease
* Severe dry eye symptoms despite having tried over a half dozen treatments

Exclusion Criteria:

* Not willing to undergo clinical trial
* Unable to comply with treatment regimen

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 3 months
  Patient Reported Outcome by Survey

SECONDARY OUTCOMES:
Visual Acuity | 3 months
  Snellen
Corneal Topography | 3 months
  Automated corneal topographic indices

CONTACTS AND LOCATIONS:
Locations (1):
- Rush Eye Associates, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: No